CLINICAL TRIAL: NCT02023268
Title: Phase III: Comparison of the Efficacy and Safety of T2762 and Vismed® in the Treatment of Moderate to Severe Dry Eye Syndrome
Brief Title: Efficacy and Safety of T2762 and Vismed® in Dry Eye Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT2762-PIII-08/13; 2013-A01292-43 (Registry Identifier: Agence Nationale de Sécurité du Médicament et des produits de santé)
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2015-11

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- T2762 (Experimental)
  Interventions: Device: T2762
- Vismed® (Active Comparator)
  Interventions: Device: Vismed®

INTERVENTIONS:
Device: T2762 — 1 drop in each eye 3 to 6 times daily during 84 days
  Arms: T2762
Device: Vismed® — 1 drop in each eye 3 to 6 times daily during 84 days
  Arms: Vismed®

SUMMARY:
Comparison of the efficacy and safety of T2762 and Vismed® in the treatment of moderate to severe Dry Eye Syndrome

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Male or female aged from ≥ 18 years old.
* Known Dry Eye Syndrome requiring artificial tears within the last 3 months prior to study selection.

Exclusion Criteria:

* Best far corrected visual acuity < 1/10
* Severe blepharitis
* Severe Dry Eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clermont-Ferrand, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T2762 | Vismed®
Started | 52 | 53
Completed | 52 | 49
Not Completed | 0 | 4
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T2762 | Vismed® | Total
Number analyzed (Participants) | 52 | 53 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 35 | 69
  >=65 years | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (12.2) | 58.5 (13.4) | 59.2 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 45 | 86
  Male | 11 | 8 | 19
Region of Enrollment [Number; unit: participants]
  France | 31 | 31 | 62
  Tunisia | 21 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Global Ocular Staining (With Oxford Scale - Ranges : 0-15)
Description: Change from Baseline in the worse eye on Day 35 (decrease of Oxford score = better outcome)
  Global Ocular Staining With the Oxford Scale measured surface damage to treated eyes(by T2762 or vismed).
Time Frame: Baseline and Day 35
Population: 14 patients with major protocol deviations were excluded of the analysed population.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- T2762: T2762: drop in each eye 3 to 6 times daily during 84 days
- Vismed: Vismed : 1 drop in each eye 3 to 6 times daily during 84 days
Arm/Group | T2762 | Vismed
Number analyzed (Participants) | 46 | 45
score on a scale | -2.5 (2.0) | -2.7 (1.7)

ADVERSE EVENTS:
Arm/Group | T2762 | Vismed®
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/53
Other Adverse Events (participants affected / at risk) | 0/52 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the results of the Trial are the sole and exclusive property of THEA, and cannot be used in whatever from without prior written agreement of THEA